CLINICAL TRIAL: NCT01774773
Title: A Single-dose Study in Healthy Japanese Male Adults to Evaluate Pharmacokinetics and Pharmacodynamics of E5501 5 mg Tablet
Brief Title: A Single-dose Study in Healthy Japanese Male Adults to Evaluate Pharmacokinetics and Pharmacodynamics of E5501 5 mg Tablet (Study E5501-J081-015)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E5501-J081-015
Record Dates: First submitted 2013-01-18; First posted 2013-01-24 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Healthy

ARMS (3):
- Group A (Experimental): E5501 5mg, then 20mg, then 40 mg, then 5mg
  Interventions: Drug: Group A: E5501 5mg, then 20mg, then 40 mg, then 5mg
- Group B (Experimental): E5501 20mg, then 40mg, then 5 mg, then 5mg
  Interventions: Drug: Group B: E5501 20mg, then 40mg, then 5 mg, then 5mg
- Group C (Experimental): E5501 40mg, then 5mg, then 20 mg, then 5mg
  Interventions: Drug: Group C: E5501 40mg, then 5mg, then 20 mg, then 5mg

INTERVENTIONS:
Drug: Group A: E5501 5mg, then 20mg, then 40 mg, then 5mg — The post-randomization phase consists of the Treatment Period 1 (Visits 2-8): participants received one 5 mg tablet under fed conditions on treatment morning for 28 days. Treatment Period II (visits 9-15): 20 mg (four 5 mg tablets) under fed conditions on treatment morning for 28 days. Treatment Period III (visits 16-22): 40 mg (eight 5 mg tablets) under fed conditions on treatment morning for 28 days.
  Treatment Period IV (visits 23-29): 5 mg tablet on treatment morning under fasted conditions for 28 days.
  The washout period of 27 days or longer was set between the administration of the study drug in Treatment Periods 1, 2 and 3 and that in Treatment Periods 2, 3 and 4 respectively.
  Arms: Group A
Drug: Group B: E5501 20mg, then 40mg, then 5 mg, then 5mg — The post-randomization phase consists of the Treatment Period 1 (Visits 2-8): participants received 20 mg (four 5 mg tablets) under fed conditions on treatment morning for 28 days. Treatment Period II (visits 9-15): 40 mg (eight 5 mg tablets) under fed conditions on treatment morning for 28 days. Treatment Period III (visits 16-22): one 5 mg tablet under fed conditions on treatment morning for 28 days.
  Treatment Period IV (visits 23-29): 5 mg tablet on treatment morning under fasted conditions for 28 days.
  The washout period of 27 days or longer was set between the administration of the study drug in Treatment Periods 1, 2 and 3 and that in Treatment Periods 2, 3 and 4 respectively.
  Arms: Group B
Drug: Group C: E5501 40mg, then 5mg, then 20 mg, then 5mg — The post-randomization phase consists of the Treatment Period 1 (Visits 2-8): participants received 40 mg (eight 5 mg tablets) under fed conditions on treatment morning for 28 days. Treatment Period II (visits 9-15): one 5 mg tablet under fed conditions on treatment morning for 28 days. Treatment Period III (visits 16-22): 20 mg (four 5 mg tablets) under fed conditions on treatment morning for 28 days.
  Treatment Period IV (visits 23-29): 5 mg tablet on treatment morning under fasted conditions for 28 days.
  The washout period of 27 days or longer was set between the administration of the study drug in Treatment Periods 1, 2 and 3 and that in Treatment Periods 2, 3 and 4 respectively.
  Arms: Group C

SUMMARY:
E5501 (5 mg, 20 mg, and 40 mg) will be administered to healthy male adults in a single-center, randomized, open-label, cross-over manner. This study will consist of 2 phases including pre-randomization (before drug administration) and postrandomization (after drug administration).

ELIGIBILITY:
Inclusion criteria;

1. Non-smokers aged 20-44 at the time of informed consent,
2. BMI is between 18.5 kg/m2 and below 25 kg/m2 at screening,
3. Platelet count is between 120,000/ microliter and below 300,000/ microliter at screening and baseline
4. Subjects and their partners can agree to use medically appropriate contraception through the study period
5. Voluntarily provided written informed consent
6. Willing and able to comply with the protocol

Exclusion criteria;

1. With a past or present history of arterial thrombosis, venous thrombosis or thrombophilia
2. With a past history of clinically significant disease within 8 weeks before study drug administration or clinically significant infection within 4 weeks before study drug administration
3. With a past surgical history that may affect the pharmacokinetics of E5501
4. Suspected to have a clinically abnormal symptom or organ dysfunction that requires treatment based on the past history, complications, subjective and objective symptoms, vital signs and body weight, electrocardiograms or clinical laboratory results at screening or baseline
5. QTcF greater than 450 ms (corrected for heart rate according to Fridericia's formula) category of the 12-lead electrocardiogram at screening or baseline

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Maximal Drug Concentration (Cmax) Under Fed Conditions | 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours post-dose
Pharmacokinetic Parameter: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] Under Fed Conditions | 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Pharmacokinetic Parameter: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - infinity)] Under Fed Conditions | 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  AUC (0 - infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Pharmacokinetic Parameter: Time to Reach Maximum Observed Plasma Concentration (Tmax) Under Fed Conditions | 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours post-dose
Pharmacokinetic Parameter: Plasma Decay Half-Life (t1/2) Under Fed Conditions | 0, 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Fuminori Ohba, Study Director — Eisai Co., Ltd.
Locations (1):
- Sumida City, Tokyo, Japan